CLINICAL TRIAL: NCT06143150
Title: Can Transthoracic Ultrasound Assessment of the Diaphragmatic Performance Predict the Outcome of Non Invasive Ventilation in Critically Ill COPD Patients With Acute Exacerbation
Brief Title: Prediction of Outcome of Non Invasive Ventilation COPD Patients by Assessment of Diaphragmatic Performance
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mona Adel, Doctor, Assiut University
Other Study IDs: Diaphragmatic performance
Record Dates: First submitted 2023-11-07; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Acute Exacerbation COPD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: transthoracic ultrasound — The following parameters will be assessed by TUS:
  Diaphragmatic copulae position and mobility (inspiratory time, excursion, diaphragmatic thickening fraction TF , excursion time E-T index )

SUMMARY:
Transthoracic ultrasonographic assessment of the diaphragmatic performance as a predictor for the outcome of NIV in critically ill COPD patients with acute exacerbation.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is considered a common disease worldwide, and it poses a major health and economic problem.

COPD was the fifth leading cause for death in 2022 and will rank third by 2030. So, it's considered a devastating disease for patients and their loved ones .

Patients presented with acute exacerbations of COPD may need respiratory intensive care unit (RICU) admission. Non invasive ventilation (NIV) is considered a cornerstone management option in patients with acute exacerbation of COPD (AECOPD). Therefore, early prediction of NIV failure may help in decision making regarding escalation to invasive mechanical ventilation To date, the diaphragm is the main respiratory muscle, and derangement of it's function is an important factor in the pathophysiology of COPD COPD patients have increased airway resistance and airflow limitation, which in turn increases the mechanical load of breathing exerted on the diaphragm Diaphragmatic weakness in COPD patients results from decreased muscle strength and mobility . Although, diaphragmatic performance is a key determinant of dyspnea in COPD patients, it is rarely assessed in clinical practice In practice, only vital sign such as respiratory rate and arterial blood gases parameters (ABG) such as PH, PaO2, PaCO2, SPO2, and fiO2/paO2 are considered predictors of NIV outcome.

Assessment of diaphragmatic function transthoracic ultrasound (TUS) is a reliable, safe and bed side method for prediction of NIV outcome . Several tools commonly applied to determine diaphragmatic function such as; fluoroscopy, Computed tomography (CT), transdiaphragmatic pressure measurement, phrenic nerve stimulation, and electromyography can't be routinely used in intensive care units due to technical challenges and limitations

ELIGIBILITY:
Inclusion Criteria:

* One Hundred fifty five critically ill COPD patients admitted to respiratory intensive care unit
* Diagnosis of COPD and COPD exacerbation is fulfilled according to GOLD 2022 criteria
* Age>40years

Exclusion Criteria:

* Age ˂ 40 years.
* Refusal to participate in the study.
* Patients with morbid obesity (BMI>40).
* Absolute indication for intubation like coma ,hemodynamic instability, or life threatening arrhythmia.
* Contraindication to NIV like untreated pneumothorax, pneumothorax with air leak, widespread facial burn or trauma, tracheotomy, or active upper gastrointestinal bleeding.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients admitted to respiratory intensive care unit with acute exacerbation
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
ultrasonographic assessement of COPD patients | Baseline
  To assess the diaphragmatic performance by transthoracic ultrasound in critically ill COPD patients with acute exacerbation

SECONDARY OUTCOMES:
Time saving | Baseline
  To estimate:
  * In hospital mortality.
  * Length of ICU stay.
  * Length of hospital stay.

REFERENCES:
- [Background] Ko FW, Chan KP, Hui DS, Goddard JR, Shaw JG, Reid DW, Yang IA. Acute exacerbation of COPD. Respirology. 2016 Oct;21(7):1152-65. doi: 10.1111/resp.12780. Epub 2016 Mar 30. PMID 27028990
- [Background] Rittayamai N, Chuaychoo B, Tscheikuna J, Dres M, Goligher EC, Brochard L. Ultrasound Evaluation of Diaphragm Force Reserve in Patients with Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2020 Oct;17(10):1222-1230. doi: 10.1513/AnnalsATS.202002-129OC. PMID 32614240
- [Background] Schulz A, Erbuth A, Boyko M, Vonderbank S, Gurleyen H, Gibis N, Bastian A. Comparison of Ultrasound Measurements for Diaphragmatic Mobility, Diaphragmatic Thickness, and Diaphragm Thickening Fraction with Each Other and with Lung Function in Patients with Chronic Obstructive Pulmonary Disease. Int J Chron Obstruct Pulmon Dis. 2022 Sep 12;17:2217-2227. doi: 10.2147/COPD.S375956. eCollection 2022. PMID 36118281
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8121160/
- See also: Related Info — https://ejmr.journals.ekb.eg/article_263842.html
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4147838/
- See also: Related Info — https://ejb.springeropen.com/articles/10.4103/ejb.ejb_99_17
- See also: Related Info — https://ouci.dntb.gov.ua/en/works/l1wn5Py7/